CLINICAL TRIAL: NCT03287960
Title: An Open Label, 1-Year Trial, Including a Double-Blind Placebo-Controlled Withdrawal Period, of Setmelanotide (RM-493), a Melanocortin 4 Receptor (MC4R) Agonist, in Leptin Receptor (LEPR) Deficiency Obesity Due to Bi-Allelic Loss-of-Function LEPR Genetic Mutation
Brief Title: Setmelanotide for the Treatment of Leptin Receptor (LEPR) Deficiency Obesity
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Rhythm Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RM-493-015; 2017-002005-36 (EudraCT Number)
Record Dates: First submitted 2017-09-14; First posted 2017-09-19 (Actual); Results first posted 2023-05-23 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: Leptin Receptor Deficiency Obesity
Keywords: LEPR deficiency obesity; setmelanotide; RM-493; Leptin receptor; Obesity; Melanocortin 4 receptor
MeSH Terms: conditions — Obesity | interventions — setmelanotide

STUDY DESIGN:
Intervention Model Description: Open-label with an 8 week Double-Blind Placebo-Controlled Withdrawal Period
Masking Description: During the 8 week double-blind placebo-controlled withdrawal period, participants received 4 weeks of daily setmelanotide and 4 weeks of daily placebo. Participants, investigators, and sites remained blinded as to when placebo treatment was administered.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Setmelanotide (Experimental): Participants received titrated doses of setmelanotide once daily, by SC injection during titration period for 2 - 12 weeks. Thereafter, participants continued setmelanotide at their specific therapeutic dose for an additional 10 weeks during the open label treatment period. Participants who achieved at least a 5 kg weight loss (or at least 5% weight loss if baseline body weight was <100 kg) at the end of the open label treatment period, continued into the 8-week double-blind withdrawal period and received 4 weeks setmelanotide and 4 weeks placebo. Following the withdrawal period, participants entered open label treatment period and received setmelanotide to complete approximately 52 weeks (~1 year) of treatment at a therapeutic dose.
  Interventions: Drug: Setmelanotide; Drug: Placebo

INTERVENTIONS:
Drug: Setmelanotide — Once daily subcutaneous injection
  Other Names: RM-493
Drug: Placebo — Once daily subcutaneous injection

SUMMARY:
To demonstrate statistically significant and clinically meaningful effects of setmelanotide on percent body weight change in participants with LEPR deficiency obesity due to rare bi-allelic or loss-of function mutations at the end of 1 year of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Bi-allelic, homozygous or compound heterozygous (a different gene mutation on each allele) genetic status for the LEPR gene, with the loss-of-function (LOF) variant for each allele conferring a severe obesity phenotype.
2. Age 6 years and above. 6+: Germany, Netherlands, UK. 12+: France
3. If adult age ≥18 years, obesity with body mass index (BMI) ≥ 30 kilograms per meters squared (kg/m^2); if child or adolescent (< 18 years of age), obesity with weight > 97th percentile for age on growth chart assessment.
4. Study participant and/or parent or guardian is able to communicate well with the investigator, to understand and comply with the requirements of the study, and is able to understand and sign the written informed consent/assent, after being informed about the study.
5. Female participants of child-bearing potential must agree to use contraception as outlined in the protocol. Female participants of non-childbearing potential, defined as surgically sterile (status post hysterectomy, bilateral oophorectomy, or bilateral tubal ligation) post-menopausal for at least 12 months (and confirmed with a screening FSH level in the post-menopausal lab range), or failure to have progressed to Tanner Stage V and/or failure to have achieved menarche, do not require contraception during the study.
6. Male participants with female partners of childbearing potential must agree to a double barrier method if they become sexually active during the study. Male participants must not donate sperm during and for 90 days following their participation in the study.

Exclusion Criteria:

1. Recent intensive (within 2 months) diet and/or exercise regimen with or without the use of weight loss agents including herbal medications, that has resulted in weight loss or weight stabilization.
2. Prior gastric bypass surgery resulting in >10% weight loss durably maintained from the baseline pre-operative weight with no evidence of weight regain.
3. Diagnosis of schizophrenia, bipolar disorder, personality disorder or other Diagnostic and Statistical Manual of Mental Disorders (DSM-III) disorders that the investigator believes will interfere significantly with study compliance.
4. A Patient Health Questionnaire-9 (PHQ-9) score of ≥ 15.
5. Any suicidal ideation of type 4 or 5 on the Columbia Suicide Severity Rating Scale (C-SSRS). Any lifetime history of a suicide attempt, or any suicidal behavior in the last month.
6. Current, severe stable restrictive or obstructive lung disease arising because of extreme obesity, evidence of significant heart failure (New York Heart Association [NYHA] Class 3 or greater), or oncologic disease, if these were severe enough to interfere with the study and/or would confound the results.
7. History of significant liver disease or liver injury, or current liver assessment for a cause of abnormal liver tests [as indicated by abnormal liver function tests, alanine transaminase (ALT), aspartate transaminase (AST), alkaline phosphatase, or serum bilirubin (> 2.0 x upper limit of normal (ULN) for any of these tests)] for an etiology other than non-alcoholic fatty liver disease (NAFLD).
8. History or presence of impaired renal function as indicated by clinically significant abnormal creatinine, blood urea nitrogen (BUN), or urinary constituents (e.g., albuminuria) or moderate to severe renal dysfunction as defined by the Cockcroft Gault equation < 30 milliliter/minute (mL/min).
9. History or close family history (parents or siblings) of skin cancer or melanoma, or participant history of ocular-cutaneous albinism.
10. Significant dermatologic findings relating to melanoma or pre-melanoma skin lesions, determined as part of a screening comprehensive skin evaluation performed by a qualified dermatologist.
11. Volunteer is, in the opinion of the study investigator, not suitable to participate in the study.
12. Participation in any clinical study with an investigational drug/device within 3 months prior to the first day of dosing.
13. Significant hypersensitivity to study drug.
14. Inability to comply with every day (QD) injection regimen.
15. Participants who have been placed in an institution through an official or court order, as well as those who are dependent on the sponsor, Investigator or study site.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2018-01-30 (Actual); Primary Completion 2020-09-25 (Actual); Study Completion 2020-09-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Meeker, MD, Study Chair — Rhythm Pharmaceuticals, Inc.
Locations (6):
- Markham Stouffville Hospital, Markham, Ontario, Canada
- Institute of Cardiometabolism and Nutrition / Pitié-Salpêtrière Hospital, Paris, France
- University of Ulm, Ulm, Germany
- Erasmus Medical Center, Rotterdam, Netherlands
- Hôpital Félix GUYON, Saint-Denis, Reunion
- University of Cambridge Metabolic Research Laboratories, Cambridge, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Clement K, van den Akker E, Argente J, Bahm A, Chung WK, Connors H, De Waele K, Farooqi IS, Gonneau-Lejeune J, Gordon G, Kohlsdorf K, Poitou C, Puder L, Swain J, Stewart M, Yuan G, Wabitsch M, Kuhnen P; Setmelanotide POMC and LEPR Phase 3 Trial Investigators. Efficacy and safety of setmelanotide, an MC4R agonist, in individuals with severe obesity due to LEPR or POMC deficiency: single-arm, open-label, multicentre, phase 3 trials. Lancet Diabetes Endocrinol. 2020 Dec;8(12):960-970. doi: 10.1016/S2213-8587(20)30364-8. Epub 2020 Oct 30. PMID 33137293

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled into the pivotal cohort (11 participants) or supplemental cohort (4 participants).
  Pivotal cohort: Set of participants under study constituted a collection of detailed clinical case reports with a comprehensive baseline and past medical history assessment and complete clinical efficacy, safety and laboratory evaluations conducted for each participant.
  Supplemental cohort: Any additional participants enrolled were included in supplemental cohort.
Pre-assignment Details: At screening, a blood sample was obtained for genotyping for mechanisms considered to be possibly related to the safety or efficacy response to the study medication (e.g., other obesity related genes). Complete physical, relevant bloodwork and other standard assessments were performed.
Groups:
- Setmelanotide: Participants received titrated doses of setmelanotide once daily, by subcutaneous (SC) injection during titration period for 2 - 12 weeks. Thereafter, participants continued setmelanotide at their specific therapeutic dose for an additional 10 weeks during the open label treatment period. Participants who achieved at least a 5 kg weight loss (or at least 5% weight loss if baseline body weight was <100 kg) at the end of the open label treatment period, continued into the 8-week double-blind withdrawal period and received 4 weeks setmelanotide and 4 weeks placebo. Following the withdrawal period, participants entered open label treatment period and received setmelanotide to complete approximately 52 weeks (~1 year) of treatment at a therapeutic dose.
Period: Titration Period (2 to 12 Weeks)
Arm/Group | Setmelanotide
Started | 15
Completed | 15
Not Completed | 0
Period: Open-Label Period (10 Weeks)
Arm/Group | Setmelanotide
Started | 15
Completed | 14
Not Completed | 1
Not completed — Adverse Event | 1
Period: Double-Blind Withdrawal Period (8 Weeks)
Arm/Group | Setmelanotide
Started | 14
Completed | 14
Not Completed | 0
Period: Open-Label Period (32 Weeks)
Arm/Group | Setmelanotide
Started | 14
Completed | 13
Not Completed | 1
Not completed — Serious Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Setmelanotide
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 5
  Between 18 and 65 years | 10
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 21.67 (8.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 13
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 12
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Count of Participants; unit: Participants]
  Netherlands | 3
  United Kingdom | 1
  France | 6
  Germany | 4
  Canada | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Reached ≥10% Weight Loss Threshold After 1 Year (Pivotal Cohort)
Description: The percentage of participants who met the ≥10% weight loss threshold (responders) after approximately Week 52 (~1 year) of treatment were analyzed.
Time Frame: Week 52
Population: The full analysis set (FAS) consisted of participants who received any of the study drug injections and at least one baseline assessment (included those who did and did not demonstrate ≥5 kg weight loss or 5% of body weight if weight is <100 kg at baseline over the initial12-week open label treatment period and proceeded into the double blind, placebo-controlled withdrawal period). Participants in pivotal cohort were included in the analysis.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Groups:
- Setmelanotide (Entire Study): Participants received setmelanotide once daily by SC injection for approximately 52 weeks (~ 1 year).
Arm/Group | Setmelanotide (Entire Study)
Number analyzed (Participants) | 11
percentage of participants | 45.5 [19.96 to 72.88]
Statistical Analysis 1: Comparison: Setmelanotide (Entire Study); Test type: Other — Two-sided confidence interval obtained using Clopper-Pearson method and one-sided p-value obtained from exact binomial test, testing that at least 5% of participants in the population of interest will achieve 10% weight loss; p = 0.0001, Clopper-Pearson method

2. Secondary Outcome: Percentage of Participants Who Reached ≥10% Weight Loss Threshold After 1 Year (Pivotal + Supplemental Cohort)
Description: as for outcome 1
Time Frame: Week 52
Population: FAS Population. Participants in pivotal and supplemental cohort were included in the analysis.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Setmelanotide (Entire Study)
Number analyzed (Participants) | 15
percentage of participants | 53.3 [30.00 to 75.63]
Statistical Analysis 1: Comparison: Setmelanotide (Entire Study); Test type: Other — Two-sided confidence interval (CI) obtained using Clopper-Pearson method and one-sided p-value obtained from exact binomial test, testing that at least 5% of patients in the population of interest would achieve 10% weight loss; p < 0.0001, Clopper-Pearson method

3. Secondary Outcome: Mean Percent Change From Baseline in Body Weight
Description: The mean percent change from baseline in body weight at 52 weeks was analyzed.
Time Frame: Baseline and Week 52
Population: The Designated Use Set (DUS) consisted of participants who received any of the study drug injections, demonstrated ≥5 kg weight loss [or 5% of body weight if weight was <100 kg at baseline] during the initial 12-week open label treatment period, and proceeded into the double-blind, placebo-controlled withdrawal period. Participants in pivotal and supplemental cohort were included in the analysis.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Setmelanotide (Entire Study)
Number analyzed (Participants) | 10
Percent change | -12.34 (7.534)
Statistical Analysis 1: Comparison: Setmelanotide (Entire Study); Test type: Other — Model based summary statistics from longitudinal mixed analysis of variance (ANOVA) model with fixed effect for visit, baseline body weight and random effect for participant, one sided p-value from model; p < .0001, ANOVA; Longitudinal mixed ANOVA; Least Squares Mean = -12.37, 90% CI 2-sided [-15.08 to -9.66]

4. Secondary Outcome: Mean Percent Change From Baseline in Hunger Score ('Most Hunger')
Description: The mean percent change in hunger scores for participants ≥12 years of age with leptin receptor (LEPR) deficiency obesity in treatment with setmelanotide was evaluated. Hunger score ranged from 0 - 10 on a Likert-type scale; 0 = not hungry at all and 10 = hungriest possible. On the Daily Hunger Questionnaire, each of the 3 items (average hunger, most/worst hunger, and morning hunger) was scored separately and averaged on a weekly basis.
Time Frame: Baseline and Week 52
Population: DUS Population. Participants in pivotal and supplemental cohort were included in the analysis.
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Setmelanotide (Entire Study)
Number analyzed (Participants) | 10
Percent Change | -42.7 (27.49)
Statistical Analysis 1: Comparison: Setmelanotide (Entire Study); Test type: Other — Model based summary statistics from longitudinal mixed analysis of variance model with fixed effect for week, baseline daily hunger score and random effect for participant, one sided p-value from model; p < .0001, ANOVA; Longitudinal mixed analysis of variance (ANOVA) model; Least Squares Mean = -42.69, 90% CI 2-sided [-56.35 to -29.02]

5. Secondary Outcome: Percentage of Participants Achieving at Least 25% Improvement in Daily Hunger From Baseline
Description: The percentage of participants (≥12 years of age) achieving a ≥25% improvement from baseline in hunger score at Week 52 (i.e., after treatment with setmelanotide for 52 weeks at the therapeutic dose) was assessed. Hunger ranged from 0 - 10 on a Likert-type scale; 0 = not hungry at all and 10 = hungriest possible. On the Daily Hunger Questionnaire, each of the 3 items (average hunger, most/worst hunger, and morning hunger) was scored separately and averaged on a weekly basis.
Time Frame: Baseline and Week 52
Population: FAS population with available data at specified time point. Participants in pivotal and supplemental cohort were included in the analysis.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Setmelanotide (Entire Study)
Number analyzed (Participants) | 14
percentage of participants | 71.4 [46.00 to 89.60]
Statistical Analysis 1: Comparison: Setmelanotide (Entire Study); Test type: Other — Two-sided CI obtained using Clopper-Pearson method and one-sided p-value obtained from exact binomial test, testing that ≥5 % of participants in the population of interest would achieve ≥25 % improvement in daily hunger score; p < .0001, Clopper-Pearson method

6. Secondary Outcome: Absolute Change From Baseline in Waist Circumference
Description: Waist circumference (cm) was measured according to the National Heart, Lung, and Blood Institute (NHLBI) criteria. Waist circumference was measured when participants were fasting at approximately the same time at each visit. The absolute change from baseline in waist circumference was assessed.
Time Frame: Baseline and Week 52
Population: DUS population with available data at specified time point. Participants in pivotal and supplemental cohort were included in the analysis.
Measure: Mean (Standard Deviation); unit: Centimeter
Arm/Group | Setmelanotide (Entire Study)
Number analyzed (Participants) | 10
Centimeter
  Baseline | 131.58 (24.047)
  Change at Week 52: number analyzed (Participants) | 7
  Change at Week 52 | -9.80 (6.095)
Statistical Analysis 1: Comparison: Setmelanotide (Entire Study); Test type: Other — Model based summary statistics from longitudinal mixed analysis of variance model with fixed effect for visit, baseline waist circumference and random effect for participant, one sided p-value from model; p = 0.0031, ANOVA; Longitudinal mixed ANOVA; Least Squares Mean = -8.9, 90% CI 2-sided [-14.10 to -3.61]

7. Secondary Outcome: Absolute Change in Body Weight (Reversal of Weight Loss) During Double-Blind Placebo-Controlled Withdrawal Period
Description: A comparison of weight change was evaluated during the 8 week placebo-controlled withdrawal period for each participant, during which each participant received 4 weeks of placebo and 4 weeks active therapy in a blinded fashion.
Time Frame: Baseline and Week 8 of withdrawal period
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Kilogram
Groups:
- Setmelanotide (Double-Blind): Participants received setmelanotide once daily by SC injection for 4 weeks and placebo matched to setmelanotide for 4 weeks during the double-blind placebo controlled withdrawal period.
Arm/Group | Setmelanotide (Double-Blind)
Number analyzed (Participants) | 9
Kilogram
  Change at Week 4: Setmelanotide | -1.2 (3.04)
  Change at Week 4: Placebo: number analyzed (Participants) | 7
  Change at Week 4: Placebo | 4.9 (2.82)

8. Secondary Outcome: Absolute Daily Hunger Reduction Score During the Double-Blind Placebo-Controlled Withdrawal Period
Description: The absolute score in daily hunger reduction during the double-blind placebo-controlled withdrawal period (≥12 Years of Age) was assessed. Hunger ranged from 0 - 10 on a Likert-type scale; 0 = not hungry at all and 10 = hungriest possible. On the Daily Hunger Questionnaire, each of the 3 items (average hunger, most/worst hunger, and morning hunger) was scored separately and averaged on a weekly basis. The weekly average hunger score of the daily worst (most) hunger score in 24 hours is the hunger score used to assess this study endpoint. Lower scores represent lower hunger, higher scores represent greater hunger.
Time Frame: Week 8 of withdrawal period
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Setmelanotide (Double-Blind)
Number analyzed (Participants) | 9
units on a scale
  Setmelanotide | 3.4 (1.63)
  Placebo: number analyzed (Participants) | 8
  Placebo | 6.3 (2.13)

9. Secondary Outcome: Mean Percent Change From Baseline in Body Mass Index
Description: The mean percent change from baseline in body mass index (BMI) was assessed.
Time Frame: Baseline and Week 52
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Setmelanotide (Entire Study)
Number analyzed (Participants) | 7
Percent change | -14.24 (9.096)
Statistical Analysis 1: Comparison: Setmelanotide (Entire Study); Test type: Other — Model based summary statistics from longitudinal mixed analysis of variance model with fixed effect for week, baseline BMI and random effect for participant, one sided p-value from model; p < .0001, ANOVA; Longitudinal mixed ANOVA model; Least Squares Mean = -14.0, 90% CI 2-sided [-16.80 to -11.20]

10. Secondary Outcome: Change From Baseline in Glucose Parameters
Description: Glucose parameters included glucose, glycated hemoglobin (HbA1c) and Oral glucose tolerance test (OGTT). Data is planned to be reported only for change from baseline in glucose levels.
Time Frame: Baseline and Week 52
Population: The Safety Analysis Set (SAS) was defined as all participants who received any study drug injections at least one post-dose safety assessment. Participants with available data were analyzed. Participants in pivotal and supplemental cohort were included in the analysis.
Measure: Mean (Standard Deviation); unit: millimole per liter
Arm/Group | Setmelanotide (Entire Study)
Number analyzed (Participants) | 15
millimole per liter
  Baseline | 5.586 (2.3740)
  Change at Week 52: number analyzed (Participants) | 6
  Change at Week 52 | -0.465 (1.4350)

ADVERSE EVENTS:
Time Frame: From first dose up to ~30 days after last dose of study drug (Up to ~ 1 year)
Description: SAS population. Participants in pivotal and supplemental cohort were included. Adverse events were analyzed for participants in placebo & setmelanotide groups combined as one group per planned analysis.
Arm/Group | Setmelanotide
All-Cause Mortality (participants affected / at risk) | 1/15
Serious Adverse Events (participants affected / at risk) | 3/15
Other Adverse Events (participants affected / at risk) | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Setmelanotide (N=15)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Road Traffic Accident (Injury, poisoning and procedural complications) | 1 (1) — Leading to event
Suicidal Ideation (Psychiatric disorders) | 1 (3)
Gastric Banding Reversal (Surgical and medical procedures) | 1 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Setmelanotide (N=15)
Flushing (Vascular disorders) | 1 (1)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (3)
Eye naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Injection site erythema (General disorders) | 11 (32)
Injection site induration (General disorders) | 7 (16)
Injection site pain (General disorders) | 7 (14)
Injection site oedema (General disorders) | 6 (13)
Injection site pruritus (General disorders) | 8 (13)
Fatigue (General disorders) | 2 (9)
Injection site bruising (General disorders) | 5 (8)
Asthenia (General disorders) | 4 (7)
Influenza like illness (General disorders) | 3 (4)
Injection site haematoma (General disorders) | 2 (3)
Injection site hypersensitivity (General disorders) | 3 (3)
Chest pain (General disorders) | 1 (2)
Malaise (General disorders) | 2 (2)
Injection site atrophy (General disorders) | 1 (1)
Injection site reaction (General disorders) | 1 (1)
Injection site urticaria (General disorders) | 1 (1)
Medical device pain (General disorders) | 1 (1)
Medical device site erythema (General disorders) | 1 (1)
Oedema (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Xerosis (General disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 4 (7)
Anxiety (Psychiatric disorders) | 3 (4)
Depression (General disorders) | 2 (4)
Depressed mood (Psychiatric disorders) | 2 (2)
Suicidal ideation (General disorders) | 1 (2)
Affect lability (General disorders) | 1 (1)
Drug abuse (Psychiatric disorders) | 1 (1)
Fear of injection (Psychiatric disorders) | 1 (1)
Illusion (Psychiatric disorders) | 1 (1)
Dysmenorrhoea (Reproductive system and breast disorders) | 1 (5)
Spontaneous penile erection (Reproductive system and breast disorders) | 4 (5)
Ejaculation disorder (Reproductive system and breast disorders) | 1 (2)
Metrorrhagia (Reproductive system and breast disorders) | 1 (2)
Amenorrhoea (Reproductive system and breast disorders) | 1 (1)
Ovarian cyst (Reproductive system and breast disorders) | 1 (1)
Vaginal haemorrhage (General disorders) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1)
Joint Injury (Injury, poisoning and procedural complications) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Blood creatine phosphokinase abnormal (Investigations) | 1 (1)
Blood follicle stimulating hormone increased (Investigations) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 1 (1)
Blood luteinising hormone increased (Investigations) | 1 (1)
Blood urea decreased (Investigations) | 1 (1)
Blood uric acid increased (Investigations) | 1 (1)
Heart rate increased (Investigations) | 1 (1)
Insulin tolerance test abnormal (Investigations) | 1 (1)
Neutrophil count increased (Investigations) | 1 (1)
Weight increased (Investigations) | 1 (1)
Cardiac flutter (Cardiac disorders) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (3)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 3 (3)
Eosinophilia (Blood and lymphatic system disorders) | 1 (3)
Iron deficiency anemia (Blood and lymphatic system disorders) | 1 (1)
Headache (Nervous system disorders) | 5 (18)
Dizziness (Nervous system disorders) | 4 (5)
Sleep paralysis (Nervous system disorders) | 1 (3)
Presyncope (Nervous system disorders) | 1 (2)
Sciatica (Nervous system disorders) | 1 (2)
Syncope (Nervous system disorders) | 1 (2)
Migraine (Nervous system disorders) | 1 (1)
Tic (Nervous system disorders) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 1 (2)
Tinnitus (Ear and labyrinth disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 8 (16)
Abdominal pain upper (Gastrointestinal disorders) | 4 (13)
Diarrhea (Gastrointestinal disorders) | 7 (13)
Constipation (Gastrointestinal disorders) | 2 (3)
Abdominal pain (Gastrointestinal disorders) | 1 (2)
Gingival discolouration (Gastrointestinal disorders) | 1 (2)
Vomiting (Gastrointestinal disorders) | 2 (2)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 1 (1)
Cholestasis (Hepatobiliary disorders) | 1 (1)
Hepatocellular injury (Hepatobiliary disorders) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1)
Renal colic (Renal and urinary disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 11 (20)
Erythema (Skin and subcutaneous tissue disorders) | 2 (3)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 (2)
Skin striae (Skin and subcutaneous tissue disorders) | 1 (2)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (2)
Hair growth rate abnormal (Skin and subcutaneous tissue disorders) | 1 (1)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1 (1)
Lentigo (Skin and subcutaneous tissue disorders) | 1 (1)
Lipodystrophy acquired (Skin and subcutaneous tissue disorders) | 1 (1)
Melanocytic naevus (Skin and subcutaneous tissue disorders) | 1 (1)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (1)
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (7)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (4)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 (3)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Torticollis (Musculoskeletal and connective tissue disorders) | 1 (1)
Hypothyroidism (Endocrine disorders) | 2 (2)
Hypogonadism (Endocrine disorders) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (2)
Dyslipidaemia (Metabolism and nutrition disorders) | 1 (1)
Folate deficiency (Metabolism and nutrition disorders) | 1 (1)
Glucose tolerance impaired (Metabolism and nutrition disorders) | 1 (1)
Gout (Metabolism and nutrition disorders) | 1 (1)
Vitamin A deficiency (Metabolism and nutrition disorders) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (6)
Nasopharyngitis (Infections and infestations) | 4 (6)
Gastrointestinal infection (Infections and infestations) | 2 (2)
Influenza (Infections and infestations) | 1 (2)
Pharyngitis (Infections and infestations) | 2 (2)
Rhinitis (Infections and infestations) | 2 (2)
Arthritis viral (Infections and infestations) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1)
Fungal infection (Infections and infestations) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1)
Injection site abscess (Infections and infestations) | 1 (1)
Otitis externa (Infections and infestations) | 1 (1)

LIMITATIONS AND CAVEATS:
Based on meetings with the Federal Drug Administration (FDA), the structure of the endpoints was slightly different in the statistical analysis plan (SAP) and the protocol.

In addition, there was no planned comparison to a randomized placebo group given the rarity of monogenic LEPR deficiency obesity.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All information regarding setmelanotide supplied by Rhythm to the investigator is privileged and confidential information. The investigator agrees to use this information to accomplish the study and will not use it for other purposes without consent from Rhythm. The information obtained from the clinical study will be used towards the development of setmelanotide and may be disclosed to regulatory authority(ies), other investigators, corporate partners, or consultants as required.

DOCUMENTS (2):
  • Study Protocol (2018-12-10): https://cdn.clinicaltrials.gov/large-docs/60/NCT03287960/Prot_000.pdf
  • Statistical Analysis Plan (2019-04-16): https://cdn.clinicaltrials.gov/large-docs/60/NCT03287960/SAP_001.pdf